CLINICAL TRIAL: NCT00870181
Title: Adenovirus-Mediated Delivery of Herpes Simplex Virus Thymidine Kinase Administration Improves Outcome of Recurrent High-Grade Glioma
Brief Title: ADV-TK Improves Outcome of Recurrent High-Grade Glioma
Acronym: HGG-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of Department of Gynecology and Obstetrics, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009HGG-01
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Glioma of Brain; Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Surgical Procedures, Operative; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADV-TK/GCV (Experimental): ADV-TK was administered via intraarterial cerebral infusion. Systemic GCV therapy was delivered at a dose of 5mg/kg intravenous, every 12 h at 36 hours after ADV-TK therapy.
  Interventions: Biological: ADV-TK/GCV
- Control group (Active Comparator): Patients received surgery or systemic chemotherapy or palliative care.
  Interventions: Procedure: Surgery; Drug: systemic chemotherapy

INTERVENTIONS:
Biological: ADV-TK/GCV — gene therapy
  Arms: ADV-TK/GCV
Procedure: Surgery
  Arms: Control group
Drug: systemic chemotherapy
  Arms: Control group

SUMMARY:
Malignant gliomas are the most common primary brain tumor in adults, but the prognosis for patients with these tumors remains poor despite advances in diagnosis and standard therapies such as surgery, radiation therapy, and chemotherapy. The advantages of ADV-TK gene therapy highlight its efficacy and safety for glioma patients. This clinical trial was conducted to assess the anti-tumor efficacy and safety of intraarterial cerebral infusion of replication-deficient adenovirus mutant ADV-TK, in combination with systemic intravenous GCV administration in patients with recurrent high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed WHO grades 3 to 4 malignant glioma
* Diagnosed recurrence or progression by clinical or radiological evidence
* Fit for intraarterial infusion and intravenous chemotherapy
* Adequate hepatic, renal, and hematologic function.
* Legal age ≥18 years
* Life expectancy ≥12 weeks
* Eastern Cooperative Oncology Group performance (ECOG) ≥2
* Chemotherapy completion ≥4 weeks prior and recovery from drug induced toxicities.

Exclusion Criteria:

* Active pregnancy
* Prior gene therapy
* Second primary tumor
* Gravidity, lactation, hypersensitivity to antiviral drugs, immunologic deficit, active uncontrolled infections
* Requiring treatment with warfarin or any other anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary end point was 6-month progression-free survival rate (PFS-6) | 6 months

SECONDARY OUTCOMES:
progression-free survival (PFS) | 3 years
overall survival (OS) | 3 years
safety | 1. at the time during treatments; 2. at 6-month; 3. at the end of 1-year following-up; 4. at the end of 2-year following up; 5. at the time the patient censored.
clinical benefit | at the end of 2nd ADK-TK/GCV therapy
  the rate of complete response, plus partial response, plus stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Ma Ding, M.D., Study Director — Tongji Hospital of HUST
Locations (1):
- Beijing YouAn Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ji N, Weng D, Liu C, Gu Z, Chen S, Guo Y, Fan Z, Wang X, Chen J, Zhao Y, Zhou J, Wang J, Ma D, Li N. Adenovirus-mediated delivery of herpes simplex virus thymidine kinase administration improves outcome of recurrent high-grade glioma. Oncotarget. 2016 Jan 26;7(4):4369-78. doi: 10.18632/oncotarget.6737. PMID 26716896